CLINICAL TRIAL: NCT03523026
Title: The Effects of Peripheral and Respiratory Muscle Training in Coronary Artery Patients With Metabolic Syndrome: A Randomized, Prospective, Double-Blind and Controlled Trial
Brief Title: The Effects of Muscle Training in Coronary Artery Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Kıymet Muammer, MSc PT, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kıymet Muammer
Record Dates: First submitted 2018-04-14; First posted 2018-05-14 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-09

CONDITIONS: Metabolic Syndrome; Coronary Artery Disease
Keywords: Metabolic Syndrome; Coronary Artery Patients; Neuromuscular Electrical Stimulation; Respiratory Muscle Training; Peripheral Muscle Training
MeSH Terms: conditions — Metabolic Syndrome; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMES and Peripheral Muscle Training (Experimental): Neuromuscular Electrical Stimulation (NMES) and Peripheral Muscle Training
  NMES frequency will be 30 Hertz and the application time will be 30 minutes.Treatment will be programmed for 3 days per week.
  Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation 3 times per week.The program will continue for 6 weeks.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Peripheral Muscle Training
- IMT and Peripheral Muscle Training (Experimental): Inspirator Muscle Training (IMT) and Peripheral Muscle Training
  IMT will be applied 7 days per week, twice a day for 15 minutes.
  Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation 3 times per week. The program will continue for 6 weeks.
  Interventions: Other: Inspirator Muscle Training; Other: Peripheral Muscle Training
- Peripheral Muscle Training (Experimental): Peripheral Muscle Training
  Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation 3 times per week.The program will continue for 6 weeks.
  Interventions: Other: Peripheral Muscle Training

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation(NMES) to rectus abdominis will be applied using 4 carbon silicon electrode. In the first sessions, patients ECG will be checked. Patients will be in semi-fowler position (30º),with their lower limbs to be in extension and upper limbs at their sides. The NMES frequency will be at 30 Hertz and the application time will be 30 minutes. Treatment will be programmed for 3 days per week. The patients will coordinate their breath (inspiration) with the contraction which will be generated by the electrical current. The program will continue for 6 weeks.
  Arms: NMES and Peripheral Muscle Training
Other: Inspirator Muscle Training — Inspirator Muscle Training(IMT) will be applied 7 days per week, twice a day for 15 minutes. The program will continue for 6 weeks duration under weekly control of the investigator.Training intensity will set at 30% of the maximum inspiratory pressure.
  Arms: IMT and Peripheral Muscle Training
Other: Peripheral Muscle Training — Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation 3 times per week.The program will continue for 6 weeks.

SUMMARY:
The aim of this study is to investigate the effects of peripheral and respiratory muscle training on respiratory muscle strength, respiratory functions, exercise capacity and quality of life in coronary artery patients with metabolic syndrome. Prospectively, randomly, double-blind, and controlled study. Stable coronary artery patients with metabolic syndrome will be included to the study from the Istanbul University Cardiology Institute clinic. Patients will be randomized into 3 groups; Neuromuscular Electrical Stimulation (NMES) and Peripheral Muscle Training Group (n: 20): 3 days per week for 6 weeks duration. Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks.Inspirator Muscle Training (IMT) and peripheral muscle training Group (n: 20): IMT will be applied 7 days per week, twice a day for 15 minutes. The program will continue for 6 weeks duration under weekly control of the investigator. Training intensity will set at 30% of the maximum inspiratory pressure.Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks. Peripheral Muscle Training Group (n: 20): Exercise will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks.Parameters will be recorded before and after training. Evaluation parameters:Demographic and anthropometric measurements, respiratory function test,respiratory muscle strength,dyspnea, peripheral muscle strength, 6 minutes walking test, physical activity, quality of life, depression, sleep quality and laboratory evaluation.

DETAILED DESCRIPTION:
Metabolic syndrome (MS) is a fatal endocrinopathy that appears with insulin resistance and is associated with systemic disorders such as abdominal obesity, glucose intolerance or diabetes mellitus, dyslipidemia, hypertension and coronary artery disease (CAD). The metabolic syndrome, which is regarded as an important public health problem in the world, shows a global increase.

Studies have showed that increased risk for cardiopulmonary disease is associated with people with metabolic syndrome. In the treatment of cardiopulmonary risk factors, therapeutic lifestyle changes and exercise are recommended in primary care strategy. Exercise training programs have been found to have positive effects on cardiopulmonary and metabolic parameters.It has been shown that respiratory functions are also adversely affected in these patients. In patients with metabolic syndrome, FEV1 and FVC were found to be influenced by decreased respiratory function and restrictive ventilation impairment.

Decreased respiratory functions and physical activity in patients with Metabolic Syndrome accompanied by multifactorial risks and complications will adversely affect quality of life. There are no studies in the literature that investigate the effects of peripheral and respiratory muscle training in patients with Metabolic Syndrome. Therefore, we aimed to investigate the effect of peripheral and respiratory muscle training on respiratory muscle strength, respiratory functions, exercise capacity and quality of life in patients with Metabolic Syndrome. This study also aimed to contribute to the international literature by applying respiratory muscle training in patients with coronary artery disease with metabolic syndrome. In addition, in clinically structured rehabilitation programs, in coronary artery disease patients with metabolic syndrome will be provided with a questioning of the importance of respiratory muscle training.

The study will be planned as prospective, randomized, double blind and controlled. Access to the patients will be provided through an archive of patient records and a screening through the online system of the outpatient clinic. Before and after the training patients' effort tests and biochemical tests will be requested. Evaluations before and after the training will be done by another physiotherapist. The study will be conducted prospectively, randomly, double-blind, and controlled. Patients will be randomized into 3 groups.

NMES and Peripheral Muscle Training Group (n: 20).

IMT and Peripheral Muscle Training Group (n: 20),

Peripheral Muscle Training Group (n = 20).

NMES and Peripheral Muscle Training Group: NMES to rectus abdominis will be applied using 4 carbon silicon electrode. In the first sessions, patients ECG will be checked. Patients will be in semi-fowler position (30º),with their lower limbs to be in extension and upper limbs at their sides. The NMES frequency will be at 30 Hertz and the application time will be 30 minutes. Treatment will be programmed for 3 days per week. The patients will coordinate their breath (inspiration) with the contraction which will be generated by the electrical current. Peripheral muscle training will also be given. Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks.

IMT and Peripheral Muscle Training Group: IMT will be applied 7 days per week, twice a day for 15 minutes. The program will continue for 6 weeks duration under weekly control of the investigator. Training intensity will set at 30% of the maximum inspiratory pressure. Peripheral muscle training will also be given. Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks.

Peripheral Muscle Training Group: Peripheral Muscle Training will be applied by elastic band and Proprioceptive Neuromuscular Facilitation three times per week for 6 weeks.

The rehabilitation program duration will be 6 weeks in all groups. Changes in parameters will be analyzed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Stable coronary artery disease with metabolic syndrome diagnosis
2. The ejection fraction(EF) = % 40 and EF >% 40,
3. Participation to the study will be in a voluntary basis

Exclusion Criteria:

1. Over 80 years,
2. EF <40% or New York Heart Association (NYHA) class III-IV
3. Chronic obstructive pulmonary disease (COPD) and respiratory tract infection,
4. Documented diagnosis of pulmonary, neurological,orthopedic, renal, hepatic, gastrointestinal, endocrine, oncologic
5. New or suspected thromboembolic events
6. Severe refractory hypertension
7. Acute myocardial infarction and pulmonary edema in the last 6 months,
8. Coronary artery revascularization attempts (percutaneous transluminal coronary angioplasty and coronary artery bypass surgery) and previous valve surgery in the last 6 months,
9. Cardiac pacemaker

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) | Baseline and 6 weeks
  Change from baseline Maximum Inspiratory Pressure (MIP) at 6 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MIP measurement is a non-invasive technique.
Maximum Expiratory Pressure (MEP) | Baseline and 6 weeks
  Change from baseline Maximum Expiratory Pressure (MEP) at 6 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The most commonly used method for evaluating respiratory muscles is MEP measurement is a non-invasive technique.
Functional capacity | Baseline and 6 weeks
  Change from baseline functional capacity test at 6 weeks. Functional capacity will be assessed by the 6 minute walking test. The test will be performed according to American Thoracic Society (ATS) criteria. Patients will be allowed to rest for 10 minutes before the test. Heart rate, blood pressure, respiratory frequency, oxygen saturation, fatigue and dyspnea perception will be recorded before and after the test. Walking distance will be calculated.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline and 6 weeks
  Change from baseline Forced Vital Capacity (FVC) in respiratory function test at 6 weeks. FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory Volume 1 second (FEV1) | Baseline and 6 weeks
  Change from baseline Forced Expiratory Volume 1 second (FEV1) in respiratory function . FEV1 will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory Volume 1 second / Forced Vital Capacity (FEV1 / FVC) | Baseline and 6 weeks
  Change from baseline FEV1 / FVC in respiratory function test at 6 weeks. FEV1 / FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Forced Expiratory flow from between 25% to 75% of Vital Capacity (FMF 25-75) | Baseline and 6 weeks
  Change from baseline Forced Expiratory flow from between 25% to 75% of Vital Capacity .
  FMF will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Peak flow rate (PEF) | Baseline and 6 weeks
  Change from baseline Peak flow rate (PEF) in respiratory function test at 6 weeks. PEF will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Dyspnea | Baseline and 6 weeks
  Change from baseline Dyspnea score of Medical Research Council (MRC) at 6 weeks.
  It will be evaluated by MRC.
Peripheral muscle strength | Baseline and 6 weeks
  Change from baseline peripheral muscle strength at 6 weeks. Lower extremity will be evaluated by 'sit to stand' test. Upper extremity will be evaluated by 'handgrip test'.
Maximal exercise capacity | Baseline and 6 weeks
  Change from baseline treadmill test at 6 weeks. It will be evaluated by treadmill test.
Physical Activity | Baseline and 6 weeks
  Change from baseline physical activity scores at 6 weeks. International Physical Activity Questionnaire (IPAQ) - Short Form (Turkish version of scale ).This questionnaire assesses, in minutes, the physical activity performed by the volunteers during the period of one week. The IPAQ considered all activities carried out by the volunteer (e.g. leisure, sport, exercise, and activities at home or in the garden). According to the responses, the volunteer is considered very active, active, irregularly active or sedentary, according to the intensity and time of the exercises practiced over the last week.
Quality of life level | Baseline and 6 weeks
  Change from baseline quality of life scores at 6 weeks. Short Form (SF-36) Health Survey (Turkish version of scale) The SF-36 is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning (10 items) social functioning (2 items) role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items). For each dimension item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Depression level | Baseline and 6 weeks
  Change from baseline depression scores at 6 weeks. Beck Depression questionnaire will be administered. The Beck Depression Questionnaire is an assessment scale that determines the risk of depression and the level of depressive symptoms and the measure of change in severity. It consists of 21 items. It provides 4 types of measurements. Each question contains 4 options. Each item gets a progressive score between 0-3 and the total score is obtained by their aggregation. The total varies from 0 to 63 points. Higher scores indicate higher depression.
Evaluation of sleep quality | Baseline and 6 weeks
  Change from baseline evaluation of sleep quality scores at 6 weeks.The Pittsburgh Sleep Quality Index (PSQI) assess sleep quality. It consists of seven subscales: subjective sleep efficiency, sleep latency, sleep duration, sleep quality, sleep disturbance, sleep medication use, and daytime dysfunction due to sleepiness. Subscales yield a score from 0 to 3 and PSQI total score of >5 is indicative of poor sleep.
Anthropometric measurements | Baseline and 6 weeks
  Change from baseline anthropometric measurements at 6 weeks. Waist, hip and abdominal circumference measurements will be assessed.The skinfold thickness will be measured with the skinfold caliper. These measurements will be made from specific measurement sites of chest, biceps, triceps, subscapular, abdominal, suprailiac, quadriceps, gastrocnemius.
Evaluation of fasting blood glucose in blood biochemistry | Baseline and 6 weeks
  Change from baseline fasting blood glucose measurements at 6 weeks. The blood glucose concentration in blood biochemistry will be assessed.
Evaluation of High Density Lipoprotein in blood biochemistry | Baseline and 6 weeks
  Change from baseline High Density Lipoprotein measurements at 6 weeks. The High Density Lipoprotein in blood biochemistry will be assessed.
Evaluation of Low Density Lipoprotein in blood biochemistry | Baseline and 6 weeks
  Change from baseline Low Density Lipoprotein measurements at 6 weeks. The Low Density Lipoprotein in blood biochemistry will be assessed.
Evaluation of triglyceride in blood biochemistry | Baseline and 6 weeks
  Change from baseline triglyceride measurements at 6 weeks. The triglyceride in blood biochemistry will be assessed.
Evaluation of C-Reactive Protein (CRP) in blood biochemistry | Baseline and 6 weeks
  Change from baseline C-Reactive Protein (CRP) measurements at 6 weeks. The C-Reactive Protein (CRP) in blood biochemistry will be assessed.
Evaluation of sedimentation in blood biochemistry | Baseline and 6 weeks
  Change from baseline sedimentation measurements at 6 weeks. The sedimentation in blood biochemistry will be assessed.
Evaluation of Antistreptolysin O (ASO) in blood biochemistry | Baseline and 6 weeks
  Change from baseline Antistreptolysin O (ASO) measurements at 6 weeks. The Antistreptolysin O (ASO) in blood biochemistry will be assessed.
Evaluation of Creatine phosphokinase (CPK) in blood biochemistry | Baseline and 6 weeks
  Change from baseline Creatine phosphokinase (CPK) measurements at 6 weeks. The Creatine phosphokinase (CPK) in blood biochemistry will be assessed.
Evaluation of Thyroid-Stimulating Hormone (TSH) in blood biochemistry | Baseline and 6 weeks
  Change from baseline Thyroid-Stimulating Hormone (TSH) measurements at 6 weeks. The Thyroid-Stimulating Hormone (TSH) in blood biochemistry will be assessed.
Evaluation of Brain Natriuretic Peptide (Pro-BNP) in blood biochemistry | Baseline and 6 weeks
  Change from baseline Brain Natriuretic Peptide (Pro-BNP) measurements at 6 weeks. The Brain Natriuretic Peptide (Pro-BNP) in blood biochemistry will be assessed.
Evaluation of complete blood count in blood biochemistry | Baseline and 6 weeks
  Change from baseline complete blood count measurements at 6 weeks. The complete blood count in blood biochemistry will be assessed.
Evaluation of ferritin in blood biochemistry | Baseline and 6 weeks
  Change from baseline ferritin measurements at 6 weeks. The ferritin in blood biochemistry will be assessed.
Evaluation of uric acid in blood biochemistry | Baseline and 6 weeks
  Change from baseline uric acid measurements at 6 weeks. The uric acid in blood biochemistry will be assessed.
Evaluation of creatinine in blood biochemistry | Baseline and 6 weeks
  Change from baseline creatinine measurements at 6 weeks. The creatinine in blood biochemistry will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kıymet Muammer, MSc PT, Principal Investigator — Istanbul University Cardiology Institute, Department of Physiotherapy and Rehabilitation; Fatma Karantay Mutluay, Professor, Study Director — Medipol University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Rengin Demir, Professor, Study Chair — Istanbul University Cardiology Institute, Department of Physiotherapy and Rehabilitation,; Alev Arat Özkan, Professor, Study Chair — Istanbul University Cardiology Institute,Catheter Laboratory
Locations (1):
- Kıymet Muammer, Istanbul, Fatih/Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Muammer K, Mutluay F, Demir R, Ozkan AA. Effects of peripheral and different inspiratory muscle training methods in coronary artery disease patients with metabolic syndrome: A randomized-controlled trial. Respir Med. 2020 Oct;172:106119. doi: 10.1016/j.rmed.2020.106119. Epub 2020 Aug 22. PMID 32877886